CLINICAL TRIAL: NCT05758584
Title: Effect of Vibrating Tourniquet and Distraction Cards on Pain and Anxiety Levels During Phlebotomy in Children
Brief Title: Effect of Vibrating Tourniquet and Distraction Cards on Pain and Anxiety in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Hümeyra Erdem, Register Nurse, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: pain_fear_anxiety...///
Record Dates: First submitted 2022-11-09; First posted 2023-03-07 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-02

CONDITIONS: Pain; Anxiety
Keywords: pain; anxiety; children; nurse; phlebotomy
MeSH Terms: conditions — Pain; Anxiety Disorders | interventions — Methods

STUDY DESIGN:
Intervention Model Description: randomized controlled study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): Vibrating tourniquet group
  Interventions: Other: Intervention
- Group 2 (Experimental): Distraction cards group
  Interventions: Other: Distraction card
- Group 3 (No Intervention): Control group

INTERVENTIONS:
Other: Intervention — Vibrating tourniquet
  Other Names: Vibrating tourniquet
  Arms: Group 1
Other: Distraction card — Distraction card
  Arms: Group 2

SUMMARY:
The aim of the study was to observe the effect of the use of vibrating tourniquet and distraction card on the pain, fear and anxiety levels felt during the blood collection process in children. The study was conducted between July 2021 and March 2022 as a randomized controlled study with totally 120 children in three groups. The 'Child and Parent Identification Form' was used for socio-demographic data about the child and the parent before phlebotomy. The 'Visual Analog Scale (VAS)', 'Child Fear Scale (CFS)' and 'Child Anxiety Scale-State Scale (ÇAS-D)' were used before, during and after the phlebotomy. Vibrating Tourniquet Group (intervention group 1) consists of a total of 40 children. Distraction Cards Group (intervention group 2) consists of a total of 40 children. Control group consists of a total of 40 children.

ELIGIBILITY:
Inclusion Criteria:

* The child is between the ages of 6-10,
* The child has no pain just before the procedure,
* The child has not taken any analgesic-effective medication in the last 6 hours,
* The child does not have a hearing problem,
* The child and the parent can speak and understand Turkish
* The child has a sufficient level of mental development to understand speech -Parent and child are willing to participate in the research.

Exclusion Criteria:

* Children who cannot be successfully drawn in the first application
* Children with oncological disease, epilepsy, migraine, or vestibular disorder.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
change on pain intensity as measured by Visual Analog Scale | "5-10 minutes before procedure", "during procedure" and "5 minutes after" blood collection process
  It is a 10 cm or 100 mm long horizontal or vertical line with anchor statements "no pain or pain at its least" at the left-most end and "unbearable pain or worst pain imaginable" at the right-most end. The VAS score is determined by measuring (in cm) the distance of the mark from the left end of the line.

SECONDARY OUTCOMES:
Score change on state anxiety level as measured by Child Anxiety Scale State Scale (ÇAS-D) | "5-10 minutes before procedure" and "5 minutes after procedure" blood collection process
  The scale is in the form of a thermometer with horizontal lines. For 10 horizontal lines, the line at the bottom of the thermometer, '0', represents the lowest anxiety level, and the line at the top of the thermometer, i.e., '10', represents the highest level of anxiety.
Score change on fear level as measured by Children's Fear Scale | "5-10 minutes before procedure" and "5 minutes after procedure" blood collection process
  These faces are showing different levels of anxiety. This face [point to the left-most face] shows no anxiety at all, this faces shows a little bit more [point to second face from left], a bit more [sweep finger along scale], right up to extreme anxiety [point to the last face on the right]. Have a look at these faces and choose the one that shows how much anxiety you felt during [the needle].

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences Turkey, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bergomi P, Scudeller L, Pintaldi S, Dal Molin A. Efficacy of Non-pharmacological Methods of Pain Management in Children Undergoing Venipuncture in a Pediatric Outpatient Clinic: A Randomized Controlled Trial of Audiovisual Distraction and External Cold and Vibration. J Pediatr Nurs. 2018 Sep-Oct;42:e66-e72. doi: 10.1016/j.pedn.2018.04.011. Epub 2018 May 1. PMID 29728296
- [Background] Bukola IM, Paula D. The Effectiveness of Distraction as Procedural Pain Management Technique in Pediatric Oncology Patients: A Meta-analysis and Systematic Review. J Pain Symptom Manage. 2017 Oct;54(4):589-600.e1. doi: 10.1016/j.jpainsymman.2017.07.006. Epub 2017 Jul 14. PMID 28712986
- [Background] Gerceker GO, Binay S, Bilsin E, Kahraman A, Yilmaz HB. Effects of Virtual Reality and External Cold and Vibration on Pain in 7- to 12-Year-Old Children During Phlebotomy: A Randomized Controlled Trial. J Perianesth Nurs. 2018 Dec;33(6):981-989. doi: 10.1016/j.jopan.2017.12.010. Epub 2018 Mar 17. PMID 29559294
- [Background] Diaz-Rodriguez M, Alcantara-Rubio L, Aguilar-Garcia D, Perez-Munoz C, Carretero-Bravo J, Puertas-Cristobal E. The Effect of Play on Pain and Anxiety in Children in the Field of Nursing: A Systematic Review. J Pediatr Nurs. 2021 Nov-Dec;61:15-22. doi: 10.1016/j.pedn.2021.02.022. Epub 2021 Mar 10. PMID 33711642